CLINICAL TRIAL: NCT07396545
Title: Effects of Ultrasound-guided External Oblique Intercostal Block Versus Erector Spinae Plane Block on Postoperative Pain in Laparoscopic Radical Gastrectomy
Brief Title: External Oblique Intercostal Block Versus Erector Spinae Plane Block on Postoperative Pain in Laparoscopic Radical Gastrectomy
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: General Hospital of Ningxia Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Lingzi-2026-1
Record Dates: First submitted 2026-02-01; First posted 2026-02-09 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Population Groups

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: On the day of surgery, after the induction of general anesthesia, the study coordinator opened the corresponding envelope in the order of recruitment. Patients were randomly assigned to receive either EOIB or ESPB, which was performed preoperatively by an experienced anesthesiologist. The anesthesiologist was aware of the intervention, but all patients, data investigator and postoperative follow-up remained blinded to group assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ESPB (Experimental): After patients entering the operating room, an intravenous line was established, and Erector Spinae Plane Block was performed under ultrasound guidance.
  Interventions: Procedure: Erector Spinae Plane Block (ESPB) group
- EOIB (Experimental): After patients entering the operating room, an intravenous line was established, and External Oblique Intercostal Plane Block was performed under ultrasound guidance.
  Interventions: Procedure: External Oblique Intercostal Plane Block

INTERVENTIONS:
Procedure: External Oblique Intercostal Plane Block — With the patient in the supine position, a high-frequency linear array probe (6-15 MHz) is used to perform a sagittal parasagittal oblique scan at the level of the 6th rib, between the right anterior axillary line and midclavicular line. The external oblique muscle, intercostal muscles, and ribs are identified. Using an in-plane technique, a 21G, 100mm block needle is inserted from a superomedial to inferolateral direction, with the needle tip positioned in the plane between the external oblique muscle and the intercostal muscles at the caudal edge of the 6th rib. 30ml of 0.375% ropivacaine is injected on each side, for a bilateral administration.
  Arms: EOIB
Procedure: Erector Spinae Plane Block (ESPB) group — With the patient in the lateral decubitus position (surgical side up), a low-frequency convex array probe (2-5 MHz) is used to perform a sagittal scan approximately 2-3 cm lateral to the spinous process of T8 or T9. The transverse process and the erector spinae muscle are identified. Using an out-of-plane technique, a 21G, 100mm block needle is advanced until contact is made with the transverse process. The needle is then withdrawn 1-2 mm to position its tip within the fascial plane deep to the erector spinae muscle and superficial to the transverse process. 30 ml of 0.375% ropivacaine is injected on each side, for a bilateral administration.
  Arms: ESPB

SUMMARY:
Postoperative pain is highly prevalent following laparoscopic radical gastrectomy. Although the erector spinae plane block (ESPB) can effectively alleviate this pain, it still has many limitations. The external oblique intercostal plane block (EOIB) is a novel nerve block technique that may provide well postoperative analgesia for upper abdominal surgery. Therefore, this study employs a non-inferiority randomized controlled trial design to verify that the analgesic effect of EOIB is not inferior to that of ESPB, thereby offering more options for regional analgesia strategies in laparoscopic radical gastrectomy.

DETAILED DESCRIPTION:
Laparoscopic radical gastrectomy (including subtotal and total gastrectomy) is the most commonly used surgical approach for gastric cancer. Although this technique is less invasive than traditional open surgery, more than 50% of patients still experience moderate to severe acute pain in the early postoperative period, making effective postoperative pain management essential. Regional nerve blockade techniques have become a key component of postoperative analgesia due to their reliable analgesic effect and significant reduction in opioid consumption.

The erector spinae plane block (ESPB) is considered a relatively safe nerve block for upper abdominal surgery analgesia. However, the spread of the local anesthetic and the resulting block effect are unpredictable. Moreover, ESPB cannot be performed with the patient in the supine position and may present technical challenges in obese patients.

The external oblique intercostal plane block (EOIB) is a recently proposed regional block technique for the upper abdomen. This block involves injecting local anesthetic into the superficial fascial plane between the external oblique muscle and the intercostal muscles, thereby blocking the anterior rami and cutaneous branches of the intercostal nerves from T6-T10, which can provide effective analgesia for upper abdominal incision areas.

Nevertheless, current research on the analgesic effect of EOIB after laparoscopic radical gastrectomy remains limited, particularly lacking high-quality, prospective, randomized controlled studies to verify whether EOIB can achieve analgesic effects comparable to those of ESPB. Therefore, this study adopts a non-inferiority randomized controlled trial design to verify that the postoperative analgesic effect of EOIB is not inferior to that of ESPB, providing more options for regional analgesia strategies in laparoscopic radical gastrectomy.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged over 18 years
* Classified as ASA I-III
* Scheduled for elective laparoscopic radical gastrectomy under general anesthesia
* Voluntarily participated and provided written informed consent.

Exclusion Criteria:

* Chronic opioid dependence or prior use of analgesic medications for >3 months;
* Inability to communicate due to severe dementia, language barriers, or terminal illness;
* History of central and/or peripheral nervous system disorders;
* Severe renal insufficiency (serum creatinine >442 μmol/L or requiring renal replacement therapy) or severe hepatic insufficiency (Child-Pugh class C);
* Allergy to local anesthetics.
* Expected to be transferred to ICU after surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 184 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2026-02-06 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Cumulative opioid consumption within 24 hours postoperatively | 24 hours after surgery
  Cumulative opioid consumption within 24 hours postoperatively. Conversion to morphine equivalent dose (mg)

SECONDARY OUTCOMES:
Pain Intensity | 2, 6, 12, 24, 48, and 72 hours postoperatively
  Pain at rest and during coughing will be assessed using the Numerical Rating Scale (NRS, 0-10) at 2, 6, 12, 24, 48, and 72 hours postoperatively.0 represents no pain, and 10 represents the most pain.
Quality of Recovery | 24,48,72 hours after surgery
  The 15-item Quality of Recovery scale (QoR-15) was used for assessment at 24, 48, and 72 hours postoperatively. The higher the score, the better the recovery quality
sleep quality | 24,48,72 hours after surgery
  Sleep quality was assessed using the Richards-Campbell Sleep Questionnaire (RCSQ) on postoperative nights.0 points represent very poor sleep, while 100 points represent very good sleep

CONTACTS AND LOCATIONS:
Overall Officials: Xinli Ni, Doctoral, Study Chair — 86-951-674-3252
Locations (1):
- General hospital of Ningxia medical university, Yinchuan, Ningxia, China

IPD SHARING:
Plan to Share IPD: No